CLINICAL TRIAL: NCT01046097
Title: Post-marketing Surveillance Study of GSK Biologicals' Pneumococcal Conjugate Vaccine, Synflorix, When Administered According to the Local Prescribing Information in Philippines
Brief Title: Post-marketing Surveillance Study With GSK Biologicals' Pneumococcal Vaccine in Healthy Infants in Philippines
Status: Terminated | Type: Observational
Why Stopped: Local authorities no longer require routine PMS studies;GSK does not believe the study would add meaningfully to the safety data already available for Synflorix
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 113381
Record Dates: First submitted 2010-01-07; First posted 2010-01-11 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-05

CONDITIONS: Infections, Streptococcal
Keywords: Pneumococcal vaccine
MeSH Terms: conditions — Streptococcal Infections | interventions — PHiD-CV vaccine

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (1):
- Synflorix Group: Subjects receiving Synflorix™ according to local Prescribing Information. Subjects were administered with Synflorix by investigators in the course of their normal clinical practice. The vaccination schedule consisted of three doses/two doses/one dose or the booster dose of 10Pn-PD-DiT to be administered as per the local PI. First dose of the vaccine could be administered to infants as early as 6 weeks of age and minimum interval between subsequent primary doses was 4 weeks.
  Interventions: Biological: Synflorix™

INTERVENTIONS:
Biological: Synflorix™ — Intramuscular administration of three doses/two doses/one dose of primary vaccination/the booster dose/ catch-up dose(s) of Synflorix according to local prescribing information.

SUMMARY:
The purpose of this post-marketing surveillance study is to evaluate the safety of Synflorix™ when administered according to the local Prescribing Information to healthy Filipino infants.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who the investigator believes that their parents/Legally Acceptable Representative(s) (LAR(s)) can and will comply with the requirements of the protocol.
* Filipino male or female subjects whose age at the first vaccination with Synflorix™ in this PMS should not be less than 6 weeks of age.
* Filipino male or female subjects who enter the PMS at the second dose should not be less than 10 weeks of age.
* Filipino male or female subjects who enter the PMS at the third dose should not be less than 14 weeks of age.
* Filipino male or female subjects who enter the PMS at the booster dose (i.e. if they have received Synflorix™ in the previous dose/s outside the PMS) should not be less than 10 months of age. The time interval between the primary vaccination and booster dose should be at least 6 months. For the booster dose, subjects who received PCV-7/-13 or Synflorix™ in their primary vaccination series will be allowed to take part in the PMS.
* Written and signed informed consent obtained from the parents/LAR(s) of the child. Where parents/LAR(s) are illiterate, the consent form will be countersigned by a witness.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.

Exclusion Criteria:

* Acute disease and/or fever at the time of vaccine administration.
* Fever is defined as temperature ≥ 37.5°C (99.5°F) on axillary, infrared or tympanic setting.
* Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of chronic condition(s) requiring treatment such as cancer or autoimmune diseases.
* Hypersensitivity to latex (found in syringe-tip cap and plunger).
* Any contraindications as stated in the Prescribing Information.

Ages: 6 Weeks to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy Filipino infants and children aged 6 weeks of age to 5 years of age who will receive Synflorix™ as a part of routine practice as per the Prescribing Information in Philippines.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-05; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Occurrence of grade 3 unsolicited adverse events. | Within 31 days (Day 0 - Day 30) after each vaccination.

SECONDARY OUTCOMES:
Occurrence of unsolicited adverse events. | During 31 days (Day 0 - Day 30) follow-up period after each vaccination/vaccine dose.
Occurrence of serious adverse events. | From the Dose 1 up to study end.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Philippines (2):
  - GSK Investigational Site, Quezon City
  - GSK Investigational Site, Santa Mesa, Manila